CLINICAL TRIAL: NCT01941225
Title: Inhaled Iloprost, Dynamic Hyperinflation, and Oxidative Stress in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Matthew Lammi, Assistant Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GM104940-50346-S
Record Dates: First submitted 2013-09-09; First posted 2013-09-13 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Pulmonary vasculature; Inhaled iloprost; Inhaled prostacyclin; Dynamic hyperinflation; Oxidative stress; Cardiopulmonary exercise testing; B-type natriuretic peptide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Nebulized normal saline. Single administration
  Interventions: Drug: Placebo
- Inhaled iloprost 5.0 mcg (Experimental): Single administration
  Interventions: Drug: Inhaled iloprost 5.0 mcg

INTERVENTIONS:
Drug: Inhaled iloprost 5.0 mcg — Single administration
  Other Names: Ventavis
  Arms: Inhaled iloprost 5.0 mcg
Drug: Placebo — Single administration
  Other Names: Nebulized normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the role of the pulmonary vasculature in the development and progression of chronic obstructive pulmonary disease (COPD). To accomplish this, an inhaled prostacyclin (iloprost) will be given to patients with COPD and changes in oxidative stress and lung volumes during exercise will be measured.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD), the 3rd leading cause of death in the US, is a progressive disorder for which new treatments are urgently needed, as existing therapies are focused primarily on symptom relief. Oxidative stress, in part arising from inducible nitric oxide synthase (iNOS) released by the pulmonary vasculature, is critical for the development and progression of COPD; a treatment strategy focused on the pulmonary vasculature is hypothesized to be beneficial in COPD patients. This will be studied with the use of an inhaled prostacyclin analogue, iloprost, which has been approved for pulmonary hypertension and investigated in small studies of COPD patients. Potential mechanisms include reductions in dynamic hyperinflation during exercise in COPD patients or improvements in oxidative stress

ELIGIBILITY:
Inclusion Criteria:

* 40 years old or older
* Physician diagnosis of chronic obstructive pulmonary disease
* 10 or more pack-year smoking history
* FEV1/FVC <0.70
* FEV1 35-80% of predicted

Exclusion Criteria:

* Acute exacerbation of COPD within the last 30 days
* Pregnant or breast-feeding
* Contraindications to cardiopulmonary exercise testing
* Known intolerance or allergy to iloprost
* On oral corticosteroids (may be included if off for 7 days prior to testing)
* Supplemental oxygen need
* Known inflammatory disease other than COPD
* Active solid organ/hematologic malignancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Dynamic hyperinflation during maximal cardiopulmonary exercise test | Acute response (exercise testing performed 30 minutes after study drug administration)
  Dynamic hyperinflation will be measured as EELV/TLC ratio (end-expiratory lung volume/total lung capacity ratio) during exercise

SECONDARY OUTCOMES:
Blood markers of oxidative stress | Acute response (measured 10 minutes, 30 minutes, 40 minutes, and 100 minutes after study drug administration)
  8-isoprostane, superoxide dismutase, catalase, nitrite, malondialdehyde
Blood markers of inflammation | Acute response (measured 10 minutes, 30 minutes, 40 minutes, and 100 minutes after study drug administration)
  IL-1 beta, IL-6, IL-8, IL-10, IL-13, IL-18, TNF-alpha
Dead space fraction | Acute response (measured every 2 minutes during exercise, starting 30 minutes after study drug administration)
B-type natriuretic peptide | Acute response (measured 30 and 40 minutes after study drug administration)
Partial pressure of oxygen | Acute response (measured 30 minutes after study drug administration and every 2 minutes during exercise)
Metabolic and gas exchange parameters during cardiopulmonary exercise test | Acute response (throughout exercise, starting 30 minutes after study drug administration)
Blood cyclic AMP levels | Acute response (measured 10 minutes, 30 minutes, 40 minutes, and 100 minutes after study drug administration)
Blood iloprost levels | Acute response (measured 10 minutes, 30 minutes, 40 minutes, and 100 minutes after study drug administration)
Exercise time and external work performed | measured during exercise test 30 minutes after study drug administration
Borg dyspnea and leg scores | During exericse (starting 30 minutes after study drug administration)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Lammi, MD, Principal Investigator — LSU Health Sciences Center
Locations (1):
- LSU Health Sciences Center, New Orleans, Louisiana, United States